CLINICAL TRIAL: NCT03757416
Title: Outcomes After Flexor Tenosynovectomy to Treat Recurrent Carpal Tunnel Syndrome: A Prospective Study
Brief Title: Flexor Tenosynovectomy to Treat Recurrent Carpal Tunnel Syndrome
Status: Terminated | Type: Observational
Why Stopped: Low enrollment; Physician practice relocating
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 15-110
Record Dates: First submitted 2018-05-03; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: recurrent; carpal tunnel release; flexor tenosynovectomy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Recurrence | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Flexor tenosynovectomy surgery: Adult patients who will be undergoing flexor tenosynovectomy for the treatment of recurrent carpal tunnel syndrome and who have already undergone primary carpal tunnel release surgery.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — If it has been determined that the patient will be undergoing flexor tenosynovectomy for the treatment of recurrent carpal tunnel syndrome, the patient will be asked to participate in this data collection study.

SUMMARY:
The purpose of this study is to collect data on the clinical and functional outcomes of surgical management for recurrent carpal tunnel syndrome (CTS) using flexor tenosynovectomy. It is hypothesized that the outcomes of patients undergoing flexor tenosynovectomy for recurrent CTS will compare favorably to published data regarding alternative types of surgeries for the same condition.

DETAILED DESCRIPTION:
Primary carpal tunnel release (CTR) is the most common surgical procedure of the hand, but reported rates of symptom recurrence are not uncommon. Many surgical techniques have been proposed and reported for management of carpal tunnel syndrome (CTS) symptom recurrence, however there is a paucity of data on flexor tenosynovectomy for management of recurrent CTS.

This study will evaluate clinical and functional outcomes using information from pre- and post-operative physical exams, surgery data, patient-reported satisfaction and symptoms, and scores on functional measures, such as the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Patient of The Plastic Surgery Group/Hayes Hand Center
* Previous diagnosis of Carpal Tunnel Syndrome
* Diagnosis of Recurrent Carpal Tunnel Syndrome
* Underwent primary carpal tunnel release
* Undergoing isolated flexor tenosynovectomy as secondary procedure

Exclusion Criteria:

* Had incomplete primary release of transverse carpal ligament
* Had documented neuroma upon re-exploration
* Had other soft tissue tumor within carpal tunnel or providing reasonable contribution to neurologic symptoms
* Experienced fracture or other traumatic injury to wrist after primary carpal tunnel release
* Diagnosis of osteomyelitis, infectious tenosynovitis or other infectious etiology to area of interest after primary procedure
* Diagnosis of rheumatoid arthritis, psoriatic arthritis, or other inflammatory arthropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of The Plastic Surgery Group/Hayes Hand Center at Erlanger Health System
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-02; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Improvement of Symptoms | one year
  'Improvement of symptoms' versus 'No change/worsening of symptoms' of carpal tunnel syndrome following flexor tenosynovectomy. Improvement vs worsening of symptoms determined by subjective physician assessment at one-year follow-up as documented through office dictation in the medical record.

SECONDARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder, and Hand) score | one year
  standard, validated patient-reported questionnaire evaluating arm/shoulder/hand function and quality of life
Patient 'satisfaction' | one year
  Determined through patient/provider interview at one-year follow-up visit: Is the patient 'satisfied' with the results after surgery? (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: D M Jemison, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga

IPD SHARING:
Plan to Share IPD: No